CLINICAL TRIAL: NCT00041327
Title: Phase II Trial Of Induction Therapy With EPOCH Chemotherapy And Maintenance Therapy With Combivir/Interferon ALPHA-2a For HTLV-1 Associated T-Cell Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Followed By Antiviral Therapy and Interferon Alfa in Treating Patients With HTLV-1-Related Adult T-Cell Leukemia/Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-033; U01CA070019 (NIH); CDR0000069469 (Other: NCI)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Lymphoma
Keywords: stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma
MeSH Terms: conditions — Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Interferon-alpha; Etoposide; Cyclophosphamide; Doxorubicin; Lamivudine; Prednisone; Vincristine; Zidovudine

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg/d
  Other Names: Neupogen
Biological: recombinant interferon alfa — 9 mU subcutaneously per day for one year
Drug: Etoposide — 50 mg/m2/day continuous 96 hr infusion, days 1-4
  Other Names: VP-16
Drug: cyclophosphamide — 750 mg/m2 IV on day 5
  Other Names: cytoxan
Drug: doxorubicin hydrochloride — 10 mg/m2/day as a continuous 96-hour infusion days 1-4
  Other Names: adriamycin
Drug: lamivudine — 150 mg bid
  Other Names: epivir
Drug: prednisone — 60 mg/m2 given orally days 1-5
  Other Names: deltasone
Drug: vincristine sulfate — 0.4 mg/m2/day as a 96-hour continuous infusion days 1-4
  Other Names: Oncovin
Drug: zidovudine — 300 mg bid
  Other Names: AZT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Antiviral therapy may kill viruses such as HTLV-1 that can cause cancer. Interferon alfa may interfere with the growth of cancer cells. Combining chemotherapy with antiviral drugs and interferon alfa may be effective in treating adult T-cell leukemia/lymphoma.

PURPOSE: Phase II trial to determine the effectiveness of combination chemotherapy followed by antiviral therapy and interferon alfa in treating patients who have adult T-cell leukemia/lymphoma caused by HTLV-1.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of etoposide, prednisone, vincristine, cyclophosphamide, and doxorubicin (EPOCH) followed by lamivudine, zidovudine, and interferon alfa, in terms of response rate, in patients with HTLV-1-associated adult T-cell leukemia/lymphoma.
* Determine the duration of response in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the effect of this regimen on markers of virus replication and expression and immune function in these patients.

OUTLINE: This is a multicenter study.

Patients receive EPOCH chemotherapy comprising etoposide, vincristine, and doxorubicin IV continuously on days 1-5, cyclophosphamide IV over 30 minutes on day 5, and oral prednisone on days 1-5. Patients also receive filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 7 and continuing until blood counts recover. Treatment repeats every 21-28 days for at least 2 courses beyond best response or for up to 6 courses in the absence of unacceptable toxicity, disease progression, or stable disease.

Beginning 1 month after completion of EPOCH, patients receive oral lamivudine and zidovudine twice daily and interferon alfa SC daily continuously for 1 year.

Patients are followed monthly for 1 year, every 2 months for 1 year, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 10-32 patients will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed HTLV-1-associated adult T-cell leukemia/lymphoma (ATLL)

  * Previously treated ATLL allowed
* CD3-positive
* Documented HTLV-1 infection by serologic assay (ELISA, Western blot)
* Measurable or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 50-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3*
* Platelet count greater than 75,000/mm^3* NOTE: *Unless cytopenia is secondary to ATLL

Hepatic:

* Transaminase less than 7 times upper limit of normal
* Bilirubin less than 2.0 mg/dL (unless secondary to hepatic infiltration with lymphoma or isolated indirect hyperbilirubinemia associated with indinavir)

Renal:

* Creatinine less than 2.0 mg/dL (unless due to lymphoma)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study completion
* No active opportunistic infection requiring acute therapy
* No untreated thyroid disease
* No autoimmune disease
* No uncontrolled significant psychiatric disease
* No other concurrent malignancy except carcinoma in situ of the cervix or non-metastatic nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 24 hours since prior hematologic growth factors

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* Concurrent chronic therapy with potentially myelosuppressive agents allowed
* Other concurrent antiretroviral therapy for HIV, hepatitis B, or hepatitis C infection (or other indication) allowed at investigator's discretion for patients receiving therapy prior to study initiation

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2002-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Efficacy | 60 days
Duration of response | 3 years
Effects on markers of virus replication and expression and immune function | 5 years
Toxicity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lee Ratner, MD, PhD, Study Chair — Washington University Siteman Cancer Center
Locations (3):
- United States (3):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri

REFERENCES:
- [Result] Ratner L, Harrington W, Feng X, Grant C, Jacobson S, Noy A, Sparano J, Lee J, Ambinder R, Campbell N, Lairmore M; AIDS Malignancy Consortium. Human T cell leukemia virus reactivation with progression of adult T-cell leukemia-lymphoma. PLoS One. 2009;4(2):e4420. doi: 10.1371/journal.pone.0004420. Epub 2009 Feb 10. PMID 19204798